CLINICAL TRIAL: NCT00436189
Title: Whole Blood Collection Protocol For Ovarian Assay Clinical Trial In Women With Ovarian Tumors
Brief Title: Assess Cancer in Ovarian Tumors With Biomarkers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciphergen Biosystems (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OVA-001-C01
Record Dates: First submitted 2007-02-13; First posted 2007-02-16 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Ovarian Tumor
Keywords: Ovarian; Cancer; Pelvic; Mass; Tumor; Adnexal; Proteomics
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Arachnodactyly | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: Blood Draw

SUMMARY:
Purpose

The OvaRI assay clinical trial is directed at evaluating a novel proteomics-based blood test. This test is for a physician to use towards differentiating benign from malignant ovarian tumors prior to surgical intervention. Tools that can better triage women with an ovarian tumor are needed. It has been shown that women with ovarian cancer who are referred to gynecologic oncologists have better outcomes. The primary objective of this study is to demonstrate that the OvaRl assay (test) improves the preoperative identification of ovarian cancer in patients with a ovarian tumor.

DETAILED DESCRIPTION:
Study Design This is a multi-center study including low and high prevalence ovarian cancer sites. The sites are representative of all institutions where potential ovarian tumor subjects will undergo a gynecological examination with radiological exam prior to surgical intervention. A blood specimen will be taken once only from enrolled subjects. This blood specimen will be used in the evaluation of the OvaRl test to identify subjects with ovarian cancer from within a population of women with a documented ovarian mass and planned surgical intervention.

Expected Total Enrollment: Up to 1000 subjects with a documented ovarian mass Study Start: February 2007

Study Details:

Study Population:

Female subjects over the age of 18 with an ovarian tumor with planned surgical intervention will be enrolled at up to 40 sites. The sites will be demographically mixed to include, for example, large and small medical centers (universities/community hospitals), small gynecology/obstetrics groups, gynecology/oncology practices, and HMO groups.

It is anticipated up to 1000 subjects will enroll. This population will exclude minors, pregnant women, or patients with a history of malignancy in the last 10 years, with the exception of a non-melanoma skin cancer.

You will only be asked to participate in this study if you have a documented mass or tumor in your ovarian area. The Ciphergen OvaR1 assay is a proteomics-based blood test that assists the physician to determine whether the documented tumor is cancer or benign (non-cancer). This is not a necessary part of your treatment. You are already scheduled to have an operation to remove this tumor, which makes you eligible for this trial. If you agree to participate you will be one of up to 1000 people to do so.

Once you are scheduled for surgery, you will be asked to provide a blood specimen once only. The blood sample will be prior to your surgery. The sample will consist of 30-50 ml of blood (about 2-3 tablespoons) drawn from a vein in your arm. The blood specimen will be processed and blood serum specimens stored, then tested with the OvaRI assay which looks at proteomic patterns indicative of cancer or non-cancer. Your serum specimens will be assigned a coded identification number to protect your privacy. Your research blood will be drawn at the time of your routine pre-operative blood work visit or at the time of surgery depending on scheduling. The only risks and potential discomforts outside of your surgery are associated with the blood draw.

The primary principal investigator in charge of this study is Frederick R. Ueland, M.D., of the University of Kentucky.

You will not receive any personal benefit from taking part in this study. However, the information obtained from your participation may potentially benefit other patients in the future by providing helpful information about proteomic patterns connected with ovarian tumors.

Subject Participation Eligibility:

Inclusion Criteria

1. Subject is female and age 18 years or older
2. Subject has a level of understanding sufficient to agree to all tests required by the protocol, must be considered reliable and must be able to cooperate with study procedures
3. Subject signs approved written informed consent prior to any study procedures being performed
4. Subject must agree to venipuncture
5. Subject has a documented ovarian tumor with planned surgical intervention

Exclusion Criteria

1. Women under age 18
2. No planned surgical intervention
3. Decline phlebotomy
4. Diagnosis of malignancy in the last 10 years, with the exception of a non-melanoma skin cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female and age 18 years or older
2. Subject has a level of understanding sufficient to agree to all tests required by the protocol, must be considered reliable and must be able to cooperate with study procedures
3. Subject signs approved written informed consent prior to any study procedures being performed
4. Subject must agree to venipuncture
5. Subject has a documented adnexal tumor with planned surgical intervention

Exclusion Criteria:

1. Women under age 18
2. No planned surgical intervention
3. Decline phlebotomy
4. Diagnosis of malignancy in the last 10 years, with the exception of a non-melanoma skin cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-04; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Proportion of actual ovarian cancer cases among OvaRl positive patients is higher than the proportion of actual ovarian cancer cases among referred patients.

SECONDARY OUTCOMES:
Evaluate OvaRl assay plus standard clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Crutcher, Study Director — Ciphergen Biosystems, Inc.; Fred Ueland, M.D., Principal Investigator — University of Kentucky; Eric Fung, M.D., Principal Investigator — CSO Ciphergen Biosystems
Locations (18):
- United States (18):
  - Clinical Research Consultants, Hoover, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Gynecologic Oncology Associates, Newport Beach, California
  - North Coast Women's Care Medical Group Inc, Vista, California
  - Farmington Obstetrics and Gynecology Group, Avon, Connecticut
  - The GYN Center for Women's Health, Waterbury, Connecticut
  - Florida Hospital Cancer Institute, Orlando, Florida
  - OB/GYN Specialists of the Palm Beaches, West Palm Beach, Florida
  - University of Kentucky - Whitney Facility, Lexington, Kentucky
  - Maine Medical Center, Scarborough, Maine
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - HWC Women's Research Center, Miamisburg, Ohio
  - Advanced Clinical Research, Medford, Oregon
  - Chattanooga Gyn-Oncology, Chattanooga, Tennessee
  - SWRCC, Austin, Texas
  - UT South Western Medical Center at Dallas, Dallas, Texas
  - Tacoma Women's Specialists, Tacoma, Washington